CLINICAL TRIAL: NCT06868719
Title: Ketone Supplementation as a Strategy to Reduce the Negative Health Effects of High Dietary Salt in Older Adults
Brief Title: Ketone Ester And Salt (KEAS) in Older Adults
Acronym: KEAS-O
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Utah (Other); University of Missouri-Columbia (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Austin Robinson, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23207b; R21AG087524 (NIH)
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Salt; Excess; Hypertension; Aging; Inflammation; Blood Pressure
Keywords: Blood Pressure; Salt; Aging; Inflammation; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blinded, randomized
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized to a condition order. A single lab member, not involved in data collection or analysis, will know condition order and contents and distribute them to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo/Placebo, then Salt/Placebo, then Salt/Ketone (Active Comparator): Participants will consume each of the supplemental interventions for 10 days (in this assigned order). On Day 10 of each interventional condition, participants will arrive at the laboratory where the investigators will assess resting blood pressure, arterial stiffness, endothelial function, renal blood flow, and submaximal exercise blood pressure reactivity. Blood will be collected to investigate inflammatory and immune responses to the dietary conditions. After a washout period, participants will consume the next assigned supplemental intervention for 10 days, and repeat the Day 10 assessments. After another washout period, participants will consume the final assigned supplemental intervention for 10 days, and again repeat the Day 10 assessments.
  Interventions: Dietary Supplement: No Salt, No β-OHB; Dietary Supplement: High Salt, No β-OHB; Dietary Supplement: High Salt, High β-OHB
- Salt/Placebo, then Salt/Ketone, then Placebo/Placebo (Active Comparator): Participants will consume each of the supplemental interventions for 10 days (in this assigned order). On day 10 of each interventional condition, participants will arrive at the laboratory where the investigators will assess resting blood pressure, arterial stiffness, endothelial function, renal blood flow, and submaximal exercise blood pressure reactivity. Blood will be collected to investigate inflammatory and immune responses to the dietary conditions. After a washout period, participants will consume the next assigned supplemental intervention for 10 days, and repeat the Day 10 assessments. After another washout period, participants will consume the final assigned supplemental intervention for 10 days, and again repeat the Day 10 assessments.
  Interventions: Dietary Supplement: No Salt, No β-OHB; Dietary Supplement: High Salt, No β-OHB; Dietary Supplement: High Salt, High β-OHB
- Salt/Ketone, then Placebo/Placebo, then Salt/Placebo (Active Comparator): Participants will consume each of the supplemental interventions for 10 days (in this assigned order). On day 10 of each interventional condition, participants will arrive at the laboratory where the investigators will assess resting blood pressure, arterial stiffness, endothelial function, renal blood flow, and submaximal exercise blood pressure reactivity. Blood will be collected to investigate inflammatory and immune responses to the dietary conditions. After a washout period, participants will consume the next assigned supplemental intervention for 10 days, and repeat the Day 10 assessments. After another washout period, participants will consume the final assigned supplemental intervention for 10 days, and again repeat the Day 10 assessments.
  Interventions: Dietary Supplement: No Salt, No β-OHB; Dietary Supplement: High Salt, No β-OHB; Dietary Supplement: High Salt, High β-OHB

INTERVENTIONS:
Dietary Supplement: No Salt, No β-OHB — Participants will consume the following for ten days. Enteric capsules will be filled with a dextrose placebo. The placebo supplement will be a β-OHB-free, taste and viscosity-matched, beverage produced by KetoneAid.
Dietary Supplement: High Salt, No β-OHB — Participants will consume the following for ten days. Enteric capsules will be filled with Morton's table salt. Sodium consumption will be normalized to caloric intake (2 mg Sodium/Calorie). The placebo supplement will be a β-OHB-free, taste and viscosity-matched, beverage produced by KetoneAid.
Dietary Supplement: High Salt, High β-OHB — Participants will consume the following for ten days. Enteric capsules will be filled with Morton's table salt. Sodium consumption will be normalized to caloric intake (2 mg Sodium/Calorie). Ketone beverage will be the β-OHB supplement produced by KetoneAid. Participants will consume 24 mL (12 grams β-OHB) of the ketone beverage three times a day (total 36 grams β-OHB).

SUMMARY:
Most Americans consume excess dietary salt based on the recommendations set by the American Heart Association and Dietary Guidelines for Americans. High dietary salt impairs blood pressure control by affecting systemic blood vessels and the kidneys. These changes contribute to excess salt consumption being associated with increased risk for chronic kidney disease and cardiovascular disease, the leading cause of death in America. Salt is particularly deleterious in older adults who are more likely to exhibit salt-sensitive hypertension. However, salt consumption remains high in the United States. Thus, there is a critical need for strategies to counteract the effects of high dietary salt as consumption is likely not going to decrease. One promising option is ketones, metabolites that are produced in the liver during prolonged exercise and very low-calorie diets. While exercise and low-calorie diets are beneficial, not many people engage in these activities. Limited evidence indicates that ketone supplements improve cardiovascular health in humans. Additionally, published rodent data indicates that ketone supplements prevent high salt-induced increases in blood pressure, blood vessel dysfunction, and kidney injury. Our human pilot data also indicates that high dietary salt reduces intrinsic ketone production, but it is unclear whether ketone supplementation confers humans' protection against high salt similar to rodents. Therefore, the investigators seek to conduct a short-term high-dietary salt study to determine whether ketone supplementation prevents high dietary salt from eliciting increased blood pressure, blood vessel dysfunction, and kidney injury/impaired blood flow. The investigators will also measure inflammatory markers in blood samples and isolate immune cells that control inflammation. Lastly, the investigators will also measure blood ketone concentration and other circulating metabolites that may be altered by high salt, which could facilitate novel therapeutic targets to combat high salt.

DETAILED DESCRIPTION:
Excess salt consumption is widespread across the United States and remains a leading risk factor for developing hypertension and cardiovascular disease (CVD). The well-documented relation between HS, hypertension, and CVD risk along with the ubiquitous HS intake in the United States demonstrate a critical need for investigation into mechanisms of salt-induced CVD; and the development of therapeutic strategies to combat the consequences of HS, particularly in at-risk populations, such as older adults. The investigators have identified the liver-derived ketone body β-hydroxybutyrate (β-OHB) as a potential target to combat the negative cardiovascular health effects of HS. Circulating β-OHB concentration typically increases in response to endurance exercise or calorie restriction, both of which also reduce blood pressure (BP) and lower CVD risk. Interestingly, chronic HS consumption suppressed endogenous hepatic β-OHB production in rats, but nutritionally upregulated hepatic β-OHB production attenuated the adverse effects of HS in the rats. Specifically, using 1,3-butanediol to increase β-OHB counteracts the adverse effects of HS on resting BP, in part by acting as a vasodilator, and attenuating inflammation. The investigators' human pilot data also indicates that HS suppresses circulating β-OHB concentration in healthy young adults. However, there is a knowledge gap regarding whether increasing β-OHB during HS intake can counteract the negative effects of HS on BP and cardiovascular health in humans. Therefore, the investigators will measure resting BP (in the lab and ambulatory), endothelial function, kidney blood flow, BP responses during and after submaximal aerobic exercise and inflammatory markers in blood and isolated immune cells (i.e., monocytes). Recognizing that HS does not increase BP in everyone, several studies consistently indicate that short-term HS ingestion (days to weeks) leads to endothelial dysfunction and exaggerated BP reactivity during submaximal exercise in humans. Importantly, endothelial dysfunction contributes to atherosclerotic cardiovascular disease. Exaggerated BP responses during aerobic exercise (i.e., BP reactivity) have prognostic value for future hypertension, coronary disease risk, and cardiovascular mortality. Apart from leading to exaggerated exercise BP reactivity, the investigators have found that HS also reduces the magnitude of post-exercise hypotension (PEH) after an acute bout of submaximal aerobic exercise in healthy adults. Importantly, the reductions in BP observed after a single bout of exercise are associated with longer-term exercise reductions in BP, suggesting that some of the benefits of aerobic exercise on BP status are the result of transient reductions in BP resulting from an acute bout of exercise. Regarding the effects of HS on the immune system and inflammation, microenvironments with elevated concentrations of sodium increase the prevalence of proinflammatory phenotypes within specific immune cell subsets. For example, HS conditions activate monocytes to produce pro-inflammatory cytokines. Thus, HS-induced immune system dysregulation may further amplify BP dysregulation and CVD risk. The investigators hypothesize that increasing circulating β-OHB concentration via ketone supplementation will counteract the negative effects of HS on these measures of cardiovascular health in older adults. Interestingly, elevating β-OHB leads to greater sodium excretion under HS conditions (indicative of restoration of plasma volume homeostasis) and restores nitric oxide-dependent vasodilation in rodents. Thus, the investigators hypothesize that ketone supplementation will improve endothelial function and BP regulation during and after exercise. Though exploratory, the investigators hypothesize that β-OHB supplementation blunts the HS-induced proinflammatory alterations in monocytes and blood samples using parallel in vitro and applied approaches.

Participants will report to the laboratory for four visits. At the first visit, consent for study participation will be obtained and participants will be screened for eligibility. Participants will then be randomly assigned to a crossover schedule for exposure to salt and ketone supplementation. Supplementation conditions include [A] Placebo capsules and Placebo beverage, [B] Salt capsules and Placebo beverage, and [C] Salt capsules and Ketone beverage. Each participant will be exposed to all three conditions, however, the order of exposure will be randomly assigned. Participants will consume their placebo/salt capsules three times per day and their placebo/ketone beverage three times per day.

Participants will consume the first assigned supplement combination for nine days prior to their first scheduled experiment visit (i.e., first experimental visit is day 10 of supplement combination #1). After a washout period, participants will consume the next randomly assigned supplement combination for nine days prior to the second scheduled experiment visit (i.e., day 10 of supplement combination #2). After another washout period, participants will consume the final randomly assigned supplement combination for nine days prior to the third scheduled experiment visit (i.e., day 10 of supplement combination #3). Participation will end after the third experimental visit has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 60-85
* Resting blood pressure no higher than 150/90
* BMI below 35 kg/m2 (or otherwise healthy)
* Free of any metabolic disease (diabetes or renal), pulmonary disorders (COPD, severe asthma, or cystic fibrosis), cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular)
* Do not have any precluding medical conditions that prevent participants from exercising (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis) or giving blood (e.g., blood thinners)

Exclusion Criteria:

* High blood pressure - greater than150/90 mmHg
* Obesity (BMI > 30 kg/m2)
* History of metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, & cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular).
* Medical issues that prevent safe exercise (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis)
* Medical issues that prevent giving blood (e.g., blood thinners).
* Current smoking, using smokeless tobacco, or vaping (within past 12 months)
* Current pregnancy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure reactivity responses | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  The investigators will measure systolic and diastolic pressure using photoplethysmography at the finger and manually measure brachial pressures. Systolic and diastolic blood pressure will be assessed at rest and during submaximal cycling exercise. Blood pressure reactivity will be expressed as a change in pressure (mmHg) from baseline to a predetermined time during the stressor.

SECONDARY OUTCOMES:
Flow mediated dilation (FMD) | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  Flow-mediated vasodilation will be assessed using continuous measures of brachial artery diameter and velocity via duplex Doppler ultrasound (Hitachi Arietta 70). The brachial artery will be imaged in the longitudinal plane proximal to the medial epicondyle using a high-frequency (10-12 MHz) linear-array probe. The ultrasound probe will be stabilized using a custom-built clamp. Shear rate (sec-1) will be calculated as [(blood flow velocity (cm*s-1) *4)/blood vessel diameter (mm)] The image will be recorded throughout a 60-s baseline, a 300-s ischemic stimulus (250 mmHg), and 180 seconds post deflation. FMD will be expressed as % dilation (final diameter-baseline diameter/baseline diameter x 100) and also normalized to the shear stimulus. Allometric scaling will be used if appropriate, including if there are baseline differences in artery diameter by race or condition.

OTHER OUTCOMES:
Pulse wave velocity | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV). A high-fidelity transducer is used to obtain the pressure waveform at the carotid pulse. Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded. PWV will be expressed as cm/s.
Pulse wave analysis | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) The sampling site is the brachial artery (upper alarm instrumented with a cuff for oscillometric sphygmomanometer). PWA will be expressed as % (calculated as augmentation pressure divided by the pulse pressure).
Passive Leg movement | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  Passive leg movement will be used assessed blood flow responses to movement. The investigators will usie continuous measures of femoral artery diameter and velocity via duplex Doppler ultrasound (Hitachi Arietta 70) to calculate blood flow at rest and with the passive lelg movement. The femoral artery will be imaged in the longitudinal plane distal to the inguinal crease using a high-frequency (10-12 MHz) linear-array probe.
  Participants will be in a seated, reclined position with the lower leg free hanging. The ultrasound probe will be positioned by a lab member and the image will be recorded throughout triplicate 60-s measurements. Another lab member will independently move the lower leg through 90º range of motion at a rate of 1 Hz.
Kidney blood velocity | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  The investigators will measure renal and segmental artery blood velocity using ultrasound-based imaging at 3.5 to 5 MHz. Blood velocity will be assessed at rest and during a cold pressor test (hand in ice-cold water for 3 minutes). Renal blood flow reactivity will be expressed as a change in velocity (cm/s) from baseline to a predetermined time during the stressor.
Inflammatory cell responses to Conditions | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  Participants' blood will be used to isolate peripheral blood mononuclear cells (PBMCs) for quantification of immune cell subsets specifically counts of monocytes and t cells.
Inflammatory cytokine responses to Conditions | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  Plasma will be used for a multiplex to measure inflammatory cytokines.
Changes in circulating reactive oxygen species | After each 10-day intervention (low salt, high salt, high salt + ketone)
  Investigators will use electron paramagnetic resonance to measure reactive oxygen species (spectra units) in whole blood samples treated with a spin probe.
Changes in blood biomarkers of plasma metabolome | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  The investigators will measure changes in the plasma metabolome, including metabolites related to energy metabolism, inflammation, and oxidative stress. Plasma samples will be collected at rest.
Changes in blood biomarkers of nitric oxide bioavailability | This measure is completed on day 10 of each 10-day intervention (low salt, high salt, high salt + ketone) over 3-4 months and values will be compared across interventions.
  The investigators will measure nitric oxide metabolites (nitrate and nitrite nanomolar concentration).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate DMDA approvals
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year after completion of the trial, indefinitely

REFERENCES:
- [Background] Babcock MC, Robinson AT, Migdal KU, Watso JC, Martens CR, Edwards DG, Pescatello LS, Farquhar WB. High Salt Intake Augments Blood Pressure Responses During Submaximal Aerobic Exercise. J Am Heart Assoc. 2020 May 18;9(10):e015633. doi: 10.1161/JAHA.120.015633. Epub 2020 May 14. PMID 32406312
- [Background] Costa TJ, Linder BA, Hester S, Fontes M, Pernomian L, Wenceslau CF, Robinson AT, McCarthy CG. The janus face of ketone bodies in hypertension. J Hypertens. 2022 Nov 1;40(11):2111-2119. doi: 10.1097/HJH.0000000000003243. Epub 2022 Aug 8. PMID 35969209
- [Background] Barnett AM, Babcock MC, Watso JC, Migdal KU, Gutierrez OM, Farquhar WB, Robinson AT. High dietary salt intake increases urinary NGAL excretion and creatinine clearance in healthy young adults. Am J Physiol Renal Physiol. 2022 Apr 1;322(4):F392-F402. doi: 10.1152/ajprenal.00240.2021. Epub 2022 Feb 14. PMID 35157527
- [Background] Chakraborty S, Galla S, Cheng X, Yeo JY, Mell B, Singh V, Yeoh B, Saha P, Mathew AV, Vijay-Kumar M, Joe B. Salt-Responsive Metabolite, beta-Hydroxybutyrate, Attenuates Hypertension. Cell Rep. 2018 Oct 16;25(3):677-689.e4. doi: 10.1016/j.celrep.2018.09.058. PMID 30332647
- [Background] McCarthy CG, Chakraborty S, Singh G, Yeoh BS, Schreckenberger ZJ, Singh A, Mell B, Bearss NR, Yang T, Cheng X, Vijay-Kumar M, Wenceslau CF, Joe B. Ketone body beta-hydroxybutyrate is an autophagy-dependent vasodilator. JCI Insight. 2021 Oct 22;6(20):e149037. doi: 10.1172/jci.insight.149037. PMID 34499623
- [Background] Wenstedt EF, Verberk SG, Kroon J, Neele AE, Baardman J, Claessen N, Pasaoglu OT, Rademaker E, Schrooten EM, Wouda RD, de Winther MP, Aten J, Vogt L, Van den Bossche J. Salt increases monocyte CCR2 expression and inflammatory responses in humans. JCI Insight. 2019 Nov 1;4(21):e130508. doi: 10.1172/jci.insight.130508. PMID 31672939